CLINICAL TRIAL: NCT02106403
Title: A Study to Evaluate the Cooling Sensation and Consumer Liking of a Skin Disinfectant Spray
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 202273; RH02332 (Other: GSK)
Record Dates: First submitted 2014-03-27; First posted 2014-04-08 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-01

CONDITIONS: Skin Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Prototype disinfectant spray formulation (Experimental): 0.13% w/w Benzalkonium Chloride (BAC) and 1% Menthone Glycerin Acetal (MGA). After wounding, the product will be held approximately 10 cm above the wounding area, and sprayed twice towards the wound
  Interventions: Other: Prototype disinfectant spray formulation
- Reference product (Active Comparator): 0.13% w/w BAC. After wounding, the product will be held approximately 10 cm above the wounding area, and sprayed twice towards the wound
  Interventions: Other: Reference product
- Negative control (Placebo Comparator): 0.9% w/v sodium chloride solution. After wounding, the product will be held approximately 10 cm above the wounding area, and sprayed twice towards the wound
  Interventions: Other: Negative control

INTERVENTIONS:
Other: Prototype disinfectant spray formulation — 0.13% w/w BAC and 1% MGA. After wounding, the product will be held approximately 10 cm above the wounding area, and sprayed twice towards the wound
  Arms: Prototype disinfectant spray formulation
Other: Reference product — 0.13% w/w BAC. After wounding, the product will be held approximately 10 cm above the wounding area, and sprayed twice towards the wound
  Arms: Reference product
Other: Negative control — 0.9% w/v sodium chloride solution. After wounding, the product will be held approximately 10 cm above the wounding area, and sprayed twice towards the wound
  Arms: Negative control

SUMMARY:
The objective of this randomised, examiner and subject blinded study is to evaluate and compare cooling performance and overall consumer liking of the prototype formulation with the currently marketed wound spray and negative control in subjects with experimental wounds. For each subject, three superficial wounds will be induced on two volar forearms, by sequential tape strippings until a glistening layer is visualized. After wounding, a randomised test product will be sprayed twice on test site, and the subject will be asked to complete a questionnaire evaluating product cooling performance and overall liking.

ELIGIBILITY:
Inclusion Criteria:

* Participants in good health with healthy and intact skin on the test area
* Age 18-60 years

Exclusion Criteria:

* Pregnancy or breast-feeding
* Allergy/Intolerance
* Participants currently taking any topical or systemic treatments that may interfere with or mask the test results
* Participants who have taken any topical anti-inflammation treatment in the application area in past 2 months
* Participants who are vulnerable to any intervention
* Damaged skin close to test site, active skin disorders, any visible skin disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Guangzhou Landproof Testing Technology Co., LTD, Guangzhou, Guangdong, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Partcipants were recruited at one clinical study site in China.
Pre-assignment Details: A total of 50 participants with 1:1 ratio of male to female were screened and 50 were randomized.
Groups:
- Sequence 1: Prototype disinfectant spray was sprayed twice on first wound, followed by Reference product twice sprayed on the second wound and subsequently Negative control was sprayed twice on the third wound. At least 30 min interval was allowed between prior and next product application.
- Sequence 2: Prototype disinfectant spray was sprayed twice on first wound, followed by Negative control sprayed twice on the second wound and subsequently Reference product was sprayed twice on the third wound. At least 30 min interval was allowed between prior and next product application.
- Sequence 3: Reference product was sprayed twice on the first wound, followed by Prototype Disinfectant Spray twice sprayed on the second wound and Negative control sprayed twice on the third wound. At least 30 min interval was allowed between prior and next product application.
- Sequence 4: Reference product was sprayed twice on the first wound, followed by Negative control sprayed twice on the second wound and subsequently prototype disinfectant spray was twice sprayed on the third wound. At least 30 min interval was allowed between prior and next product application.
- Sequence 5: Negative control was sprayed twice on the first wound, followed by Prototype Disinfectant Spray twice sprayed on the second wound and Reference product sprayed twice on the third wound. At least 30 min interval was allowed between prior and next product application.
- Sequence 6: Negative control was sprayed twice on the first wound, followed by Reference product sprayed twice on the second wound and Prototype Disinfectant Spray twice sprayed on the third wound. At least 30 min interval was allowed between prior and next product application.
Period: Visit 1, Treatment Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 8 | 8 | 9 | 8 | 8 | 9
Completed | 8 | 8 | 9 | 8 | 8 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Visit 1, Treatment Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 8 | 8 | 9 | 8 | 8 | 9
Completed | 8 | 8 | 9 | 8 | 8 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Visit 1, Treatment Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 8 | 8 | 9 | 8 | 8 | 9
Completed | 8 | 8 | 9 | 8 | 8 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Follow-Up Visit 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 8 | 8 | 9 | 8 | 8 | 9
Completed | 8 | 8 | 9 | 8 | 8 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Follow-Up Visit 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 8 | 8 | 9 | 8 | 8 | 9
Completed | 8 | 8 | 9 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other Reason | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants were evaluated for baseline characteristics
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.0 (12.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Participant-perceived Cooling Sensation Immediately Post Product Application
Description: The cooling sensation was assessed immediately after the study product application on 100 millimeter (mm) Visual Analogue Scale (VAS) (0-100 mm, where 0= no cooling and 100= extreme cooling).
Time Frame: Immediately after product application
Population: Efficacy analysis was based on intent-to-treat (ITT) population defined as all randomized participants who received the product at least once and provided at least one post product use assessment of efficacy. One participant had one efficacy assessment outside the required time window but was included in ITT population
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Groups:
- Prototype Disinfectant Spray Formulation: 0.13% w/w Benzalkonium Chloride (BAC) and 1% Menthone Glycerin Acetal (MGA). After wounding, the product was held approximately 10 cm above the wounded area, and sprayed twice towards the wound.
- Reference Product: 0.13% w/w BAC. After wounding, the product was held approximately 10 cm above the wounded area, and sprayed twice towards the wound.
- Negative Control: 0.9% w/v Sodium Chloride solution. After wounding, the product was held approximately 10 cm above the wounded area, and sprayed twice towards the wound.
Arm/Group | Prototype Disinfectant Spray Formulation | Reference Product | Negative Control
Number analyzed (Participants) | 50 | 50 | 50
Score on a scale | 30.63 (4.345) | 30.15 (4.345) | 25.16 (4.345)
Statistical Analysis 1: Comparison: Prototype Disinfectant Spray Formulation vs Negative Control; The null and alternative hypotheses were: H0: product difference was null vs. Ha: product difference was not null; Test type: Superiority or Other; p = 0.0659, ANOVA; Calculated from mixed effect ANOVA analysis with treatment and assessment site as fixed effects and subject as random effect; Mean Difference (Net) = 5.46, 95% CI 2-sided [-0.37 to 11.29] — Difference was calculated as the prototype disinfectant spray formulation minus negative control such that a positive difference showed improved cooling in the prototype disinfectant spray formulation
Statistical Analysis 2: Comparison: Reference Product vs Negative Control; The null and alternative hypotheses were: H0: product difference was null vs. Ha: product difference was not null; Test type: Superiority or Other; p = 0.0928, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 4.99, 95% CI 2-sided [-0.84 to 10.81] — Difference was calculated as the reference product minus negative control such that a positive difference showed improved cooling in the reference product
Statistical Analysis 3: Comparison: Prototype Disinfectant Spray Formulation vs Reference Product; The null and alternative hypotheses were: H0: product difference was null vs. Ha: product difference was not null; Test type: Superiority or Other; p = 0.8711, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.48, 95% CI 2-sided [-5.35 to 6.31] — Difference was calculated as the prototype disinfectant spray formulation minus reference product such that a positive difference showed improved cooling in the prototype disinfectant spray formulation

2. Primary Outcome: Participant-perceived Cooling Sensation at 3 Min
Description: The cooling sensation was assessed on VAS (0-100 mm, where 0= no cooling and 100= extreme cooling) at 3 min post study product application.
Time Frame: At 3 min after product application
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Groups:
- Prototype Disinfectant Spray Formulation: 0.13% w/w BAC and 1% MGA. After wounding, the product was held approximately 10 cm above the wounded area, and sprayed twice towards the wound.
Arm/Group | Prototype Disinfectant Spray Formulation | Reference Product | Negative Control
Number analyzed (Participants) | 50 | 50 | 50
Score on a scale | 39.15 (3.726) | 29.42 (3.726) | 27.73 (3.726)
Statistical Analysis 1: Comparison: Prototype Disinfectant Spray Formulation vs Negative Control; The null and alternative hypotheses were: H0: product difference was null vs. Ha: product difference was not null; Test type: Superiority or Other; p = 0.0016, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 11.43, 95% CI 2-sided [4.43 to 18.42] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Reference Product vs Negative Control; The null and alternative hypotheses were: H0: product difference was null vs. Ha: product difference was not null; Test type: Superiority or Other; p = 0.6323, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.69, 95% CI 2-sided [-5.31 to 8.69] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Prototype Disinfectant Spray Formulation vs Reference Product; The null and alternative hypotheses were: H0: product difference was null vs. Ha: product difference was not null; Test type: Superiority or Other; p = 0.0069, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 9.73, 95% CI 2-sided [2.74 to 16.73] — [estimate comment as in outcome 1, analysis 3]

3. Primary Outcome: Participant-perceived Cooling Sensation at 5 Min
Description: The cooling sensation was assessed on VAS (0-100 mm, where 0= no cooling and 100= extreme cooling) at 5 min post study product application.
Time Frame: At 5 min after product application
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Prototype Disinfectant Spray Formulation | Reference Product | Negative Control
Number analyzed (Participants) | 50 | 50 | 50
Score on a scale | 34.46 (3.147) | 20.14 (3.147) | 22.32 (3.147)
Statistical Analysis 1: Comparison: Prototype Disinfectant Spray Formulation vs Negative Control; The null and alternative hypotheses were: H0: product difference was null vs. Ha: product difference was not null; Test type: Superiority or Other; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 12.13, 95% CI 2-sided [6.23 to 18.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Reference Product vs Negative Control; The null and alternative hypotheses were: H0: product difference was null vs. Ha: product difference was not null; Test type: Superiority or Other; p = 0.4645, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -2.18, 95% CI 2-sided [-8.09 to 3.72] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Prototype Disinfectant Spray Formulation vs Reference Product; The null and alternative hypotheses were: H0: product difference was null vs. Ha: product difference was not null; Test type: Superiority or Other; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 14.32, 95% CI 2-sided [8.41 to 20.22] — [estimate comment as in outcome 1, analysis 3]

4. Primary Outcome: Participant-perceived Cooling Sensation at 15 Min
Description: The cooling sensation was assessed on VAS (0-100 mm, where 0= no cooling and 100= extreme cooling) at 15 min post study product application.
Time Frame: At 15 min after product application
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Prototype Disinfectant Spray Formulation | Reference Product | Negative Control
Number analyzed (Participants) | 50 | 50 | 50
Score on a scale | 16.84 (2.725) | 12.45 (2.725) | 10.43 (2.725)
Statistical Analysis 1: Comparison: Prototype Disinfectant Spray Formulation vs Negative Control; The null and alternative hypotheses were: H0: product difference was null vs. Ha: product difference was not null; Test type: Superiority or Other; p = 0.0357, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 6.41, 95% CI 2-sided [0.44 to 12.38] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Reference Product vs Negative Control; The null and alternative hypotheses were: H0: product difference was null vs. Ha: product difference was not null; Test type: Superiority or Other; p = 0.5030, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 2.02, 95% CI 2-sided [-3.95 to 8.00] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Prototype Disinfectant Spray Formulation vs Reference Product; The null and alternative hypotheses were: H0: product difference was null vs. Ha: product difference was not null; Test type: Superiority or Other; p = 0.1482, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 4.39, 95% CI 2-sided [-1.59 to 10.36] — [estimate comment as in outcome 1, analysis 3]

5. Secondary Outcome: Overall Sensory Liking of Study Products
Description: Overall sensory liking of the study products was assessed immediately, 3min, 5 min and 15 min after products application. The assessment was done on a 9 point categorical scale where 1= Dislike it extremely, 2= Dislike it very much, 3= Dislike it moderately, 4= Dislike it slightly, 5= Neither like it nor dislike it, 6= Like it slightly, 7= Like it moderately, 8= Like it very much, 9= Like it extremely.
Time Frame: Immediatey, 3 min, 5 min and 15 min after product application
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Prototype Disinfectant Spray Formulation | Reference Product | Negative Control
Number analyzed (Participants) | 50 | 50 | 50
Score on a scale | 6.60 (0.199) | 6.38 (0.199) | 6.22 (0.199)

ADVERSE EVENTS:
Time Frame: AEs were collected from the start of the investigational product, and until last visit (7 days following last administration of the investigational product).
Arm/Group | Prototype Disinfectant Spray Formulation | Reference Product | Negative Control
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 1/50 | 1/50 | 1/50
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prototype Disinfectant Spray Formulation (N=50) | Reference Product (N=50) | Negative Control (N=50)
Itch in all three wounds(Wound Complication) (Injury, poisoning and procedural complications) | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.